CLINICAL TRIAL: NCT06097455
Title: First in Human, Pilot, Open-label, Prospective, Multicentre, Non-randomised Clinical Trial to Evaluate the Safety and Efficacy of ARI0003 (CART CD19/ CD269 Cells) in Patients With Relapsed/Refractory B-cell Aggressive Lymphoma
Brief Title: First in Human Study of the Infusion of ARI0003 Cells in Relapsed/Refractory to Treatment B-cell Aggressive Lymphoma
Acronym: CARTD-BG-1
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARTD-BG-1; 2023-5072-13-97-00 (Other: EU CT)
Record Dates: First submitted 2023-10-09; First posted 2023-10-24 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Refractory Non-Hodgkin Lymphoma; Relapsed Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARI0003 (Experimental): ARI0003 will be administered intravenously under a split regime. A total dose between 0.5 and 5 x106 cell/Kg will be administered in 3 administrations (fractions):
  Interventions: Genetic: ARI0003

INTERVENTIONS:
Genetic: ARI0003 — Treatment with ARI0003 cells
  Other Names: Adult autologous differentiated T-cells from peripheral blood, expanded and co-transduced lentiviruses: one containing a chimeric antigen receptor anti-CD19 and another containing an anti-CD269 (BCMA)

SUMMARY:
ths study consist in testing a CAR T therapy (ARI0003 cells (antiCD19 and antiBCMA) in patients suffering relapsed NHL (that means that symptoms of NHL reappeared ) or refractory (that means that they did not respond to other treatments). This is a first in human study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosis of CD19+ or CD269+ relapsed/refractory (R/R) aggressive B-cell lymphoma in one of the following circumstances:

  * Burkitt's lymphoma;
  * Histology not covered by approved CART19-cell products (plasmablastic lymphoma, primary effusion lymphoma, intravascular lymphoma, transformed lymphoma from marginal zone lymphoma or chronic lymphocytic leukaemia, primary cutaneous DLBCL, T-cell rich DLBCL, high-grade B-cell lymphoma, grey zone lymphoma or grade 3b follicular lymphoma); or
  * Aggressive B-cell lymphoma that is refractory or relapsing after treatment with CART19-cell therapy.

    2. Age older than 18 years. 3. ECOG performance status of 0-2. 4. Estimated life expectancy of at least 3 months. 5. Adequate venous access and absence of contraindications for lymphapheresis. 6. Signature of informed consent. 7. In patients who have received any anti-CD19 or anti-CD269 therapy (e.g. tisagenlecleucel, axicabtagene autoleucel, tafasitamab, loncastuximab, belantamab mafodotin, idecabtagene vicleucel, etc.), a centralised tumour sample confirming the expression of at least one of the antigens (either CD19 or CD269) will be needed at study inclusion

Exclusion Criteria:

* 1. Any experimental or non-commercialized therapy in the previous 4 weeks. 2. Any other concomitant neoplasia, unless it has been in complete remission for 3 years or longer, except for non-melanoma skin cancer or completely resected in situ carcinoma.

  3. Active immunosuppressive therapy except for prednisone 10 mg/day (or equivalent).

  4. Active infection requiring systemic medical therapy. 5. Active HBV or HCV infection. 6. Positive serology for HIV. 7. Any concomitant and uncontrolled medical disease. 8. Severe organic impairment defined by cardiac ejection fraction <40%, DLCO <40%, GFR <30 ml/min or bilirubin >3 times the upper limit of normality (unless due to Gilbert's syndrome).

  9. Lactating or pregnant women. 10. Men or women of childbearing potential unable or unwilling to use highly efficient contraceptive measures from the beginning until the end of the study.

  11. CNS disease in the form of a macroscopic solid lesion in the encephalon or spinal cord (isolated meningeal disease is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Rate of > grade 3 CRS and/or ICANS | in the first 30 days after ARI0003 administration
  Rate of patients who develop grade > 3 cytokine release syndrome (CRS) and/or grade > 3 immune cell associated neurotoxicity syndrome (ICANS) according to the criteria and grading defined in the international consensus document of the American Society for Transplantation and Cellular Therapy (ASTCT criteria). ASTCT score can be between 1 and 4 (being 1 the minimum value and 4 the maximum) and where higher score means worse outcome.
ORR | within 3 months post ARI0003 infusion
  Overall response rate (ORR) according to Lugano criteria (best response within 3 months post ARI0003 infusion

SECONDARY OUTCOMES:
Procedure-related mortality (PRM) | through study completion, an average of 24 months
  Procedure-related mortality (PRM), defined as any death not directly cause by the lymphoma that is related with the procedure. For the estimation of PRM, disease relapse will be considered as a competing event
Toxicity: incidence of AE | at 3 and 12 months
  Toxicity defined as the incidence of grade >3 adverse events (AEs) as per CTCAE version 5.0. The following AEs will be considered AEs of special interest (AESI): CRS, ICANS, macrophagic activation syndrome (MAS), tumour lysis syndrome (TLS), prolonged cytopenia (beyond 6 months), infections and second primary malignancies
Complete response rate | at 3 months
  Complete response rate
Duration of response, | from month 3 to study completion, an average of 24 months
  Duration of response, calculated from the time of first disease evaluation (3 months);
Progression-free survival | through study completion, an average of 24 months
  Progression-free survival, calculated from ARI-0003 cell infusion
Overall survival | through study completion, an average of 24 months
  Overall survival, calculated from ARI-0003 cell infusion

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (7):
  - CHU Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital Clínic Barcelona, Barcelona
  - H. Ramon y Cajal, Madrid
  - H.U. Virgen de la Arrixaca, Murcia
  - Hospital Central de Asturias, Oviedo
  - Hospital Son Espases, Palma de Mallorca
  - H. Clínico de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bachiller M, Barcelo-Genestar N, Rodriguez-Garcia A, Alserawan L, Dobano-Lopez C, Gimenez-Alejandre M, Castellsague J, Colell S, Otero-Mateo M, Antonana-Vildosola A, Espanol-Rego M, Ferruz N, Pascal M, Martin-Antonio B, Anguela XM, Fillat C, Olesti E, Calvo G, Juan M, Delgado J, Perez-Galan P, Urbano-Ispizua A, Guedan S. ARI0003: Co-transduced CD19/BCMA dual-targeting CAR-T cells for the treatment of non-Hodgkin lymphoma. Mol Ther. 2025 Jan 8;33(1):317-335. doi: 10.1016/j.ymthe.2024.11.028. Epub 2024 Nov 19. PMID 39563035